CLINICAL TRIAL: NCT00373906
Title: Phase II Trial pf Bortezomib in Patients With Advanced or Relapsed Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT) Type
Brief Title: Velcade in MALT Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Velcade-MALT-Lymphoma; Eudract No 2005-003077-25
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2008-05

CONDITIONS: MALT Lymphoma
Keywords: MALT Lymphoma, Bortezomib
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib (Velcade)

SUMMARY:
Bortezomib for treatment of disseminated MALT lymphoma or at relapse following HP -eradication,or chemotherapy or radiation.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the effectivity and the safety of bortezomib in patients with disseminated MALT lymphoma or at relapse following HP-eradication, or chemotherapy or radiation.

It is a phase II prospective single arm study with a target sample of 16 patients. 1.5mg/m2 Bortezomib is given intravenously on day 1,4,8,11 every three week, for a maximum of 8cycles.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically confirmed MALT lymphoma with measurable disease (stage I-IV)
* with first or greater relapse after HP-eradication, radiation or chemotherapy ,
* age > 18 years
* must be able to tolerate therapy and have adequate cardiac, renal and hepatic function
* ECOG status of <_ 2
* must be capable of understanding the purpose of the study and given written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)

PRIMARY OUTCOMES:
to evaluate the clinical potential of bortezomib
to induce objective/histologic responses in patients with MALT-Lymphoma

SECONDARY OUTCOMES:
to evaluate the impact of bortezomib on progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Markus Raderer, Prof, Principal Investigator — Department of Internal Medicine I

REFERENCES:
- [Derived] Troch M, Jonak C, Mullauer L, Puspok A, Formanek M, Hauff W, Zielinski CC, Chott A, Raderer M. A phase II study of bortezomib in patients with MALT lymphoma. Haematologica. 2009 May;94(5):738-42. doi: 10.3324/haematol.2008.001537. Epub 2009 Mar 31. PMID 19336742